CLINICAL TRIAL: NCT02704611
Title: Direct Current Stimulation Versus Sham for Treatment of Fibromyalgia: a Double Blinded Randomized Controlled Trial
Brief Title: Direct Current Stimulation for Treatment of Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dina Hatem Elhammady (Other)
Responsible Party: Sponsor-Investigator, Dina Hatem Elhammady, Clinical Professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCS in fibromyalgia
Record Dates: First submitted 2016-03-04; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2015-10

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Active Comparator): Real tDCS (2mA for 25 minutes on 5 consecutive days/week for 2 weeks with the anode centered over M1 bilaterally. Anodal tDCS for 20 minutes at 1.5mA (15 s ramp in and 15 s ramp out) will be applied daily for 10 consecutive days (5 sessions/week).
  Interventions: Device: Real tDCS
- Group II (Sham Comparator): Sham tDCS will be applied using the above described parameters in group. For sham tDCS, the placement of the electrodes, current intensity, and ramp time was identical to real tDCS stimulation group; however, the stimulation lasted only for 30 Sec.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Real tDCS — Real tDCS (2mA for 25 minutes on 5 consecutive days/week for 2 weeks with the anode centered over M1 bilaterally. Anodal tDCS for 20 minutes at 1.5mA (15 s ramp in and 15 s ramp out) will be applied daily for 10 consecutive days (5 sessions/week). The anodal electrode 24 cm² with current density of 0.08 mA (2mA/24 cm²) will be placed over the left primary motor area in group I, and the reference electrode (24 cm² will be fixed over the contralateral arm (extracephalic).
  Other Names: Real trans-cranial direct current stimulation
  Arms: Group I
Device: Sham tDCS — Sham tDCS will be applied using the above described parameters in group. For sham tDCS, the placement of the electrodes, current intensity, and ramp time was identical to real tDCS stimulation group; however, the stimulation lasted only for 30 Sec. However, since none of the patients have been experienced tDCS previously, they were unaware of which stimulation is real and which sham is. The investigator responsible for delivering tDCS had no contact with the patients.
  Other Names: Sham trans-cranial direct current stimulation
  Arms: Group II

SUMMARY:
The aim of this study is to assess the effectiveness of transcranial direct current stimulation (tDCS) in treating fibromyalgia.

Participants will be randomly assigned to one of the two groups: Group I (Intervention group) tDCS (2mA for 25 minutes on 5 consecutive days/week for 2 weeks with the anode centered over M1 bilaterally Anodal tDCS for 20 minutes at 1.5 mA (15 s ramp in and 15 s ramp out) will be applied daily for 10 consecutive days (5 sessions/week) . The anodal electrode (24 cm² with current density of 0.08 mA (2mA/24 cm²) will be placed over the left primary motor area in group I, and the reference electrode (24 cm² will be fixed over the contralateral arm (extracephalic).

Daily tDCS was given to prolong and stabilize these long-lasting after-effects. Group II will receive sham tDCS will be applied using the above described parameters in group I. For sham tDCS, the placement of the electrodes, current intensity, and ramp time was identical to real tDCS stimulation group; however, the stimulation lasted only for 30 Sec. However, since none of the patients have been experienced tDCS previously, they were unaware of which stimulation is real and which sham is. The investigator responsible for delivering tDCS had no contact with the patients. All study participants will be followed up by the same evaluation sheet and by an evaluator who are blinded to the type of intervention she /he has received.Evaluation will be done pre assessment, post 5 sessions, post 10 sessions, post one month and post 2 months by using wide spread pain index (WPI) & symptoms severity of fibromyalgia, measuring visual analogue scale (VAS), Depression and anxiety will be assessed using Hamilton Depression Scale (HDS) and anxiety scale, pain sensitivity threshold by using Electronic Von Frey unit EVF4 . Determination of human beta-endorphin level before start sessions and after end 10 sessions.

DETAILED DESCRIPTION:
The purpose of this study is to assess the effectiveness of transcranial direct current stimulation (tDCS) in relieving pain of patients with fibromyalgia. Eligible participants will be randomly assigned to one of the two groups: Group I (Intervention group) tDCS (2mA for 25 minutes on 5 consecutive days/week for 2 weeks with the anode centered over M1 bilaterally Anodal tDCS for 20 minutes at 1.5 mA (15 s ramp in and 15 s ramp out) will be applied daily for 10 consecutive days (5 sessions/week) . The anodal electrode (24 cm² with current density of 0.08 mA (2mA/24 cm²) will be placed over the left primary motor area in group I, and the reference electrode (24 cm² will be fixed over the contralateral arm (extracephalic).

Because brief exposure to tDCS has no after-effects whereas researchers used 20min duration in order to produce robust after-effects. Daily tDCS was given to prolong and stabilize these long-lasting after-effects. Group II will receive sham tDCS will be applied using the above described parameters in group I. For sham tDCS, the placement of the electrodes, current intensity, and ramp time was identical to real tDCS stimulation group; however, the stimulation lasted only for 30 Sec. However, since none of the patients have been experienced tDCS previously, they were unaware of which stimulation is real and which sham is. The investigator responsible for delivering tDCS had no contact with the patients. All study participants will be followed up by the same evaluation sheet and by an evaluator who are blinded to the type of intervention she /he has received.Evaluation will be done pre assessment, post 5 sessions, post 10 sessions, post one month and post 2 months by using wide spread pain index (WPI) & symptoms severity of fibromyalgia, measuring visual analogue scale (VAS), Depression and anxiety will be assessed using Hamilton Depression Scale (HDS) and anxiety scale, pain sensitivity threshold by using Electronic Von Frey unit EVF4 . Determination of human beta-endorphin level before start sessions and after end 10 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as fibromyalgia according to the American college of rheumatology classification, (ACR) 2010 and referred to any of the above clinics for treatment.

  * Patients must have a mean pain score ≥ 4 on a 10-point visual analog scale (VAS) during the 2 weeks preceding the clinical trial.
  * Patients from nearby districts to ensure good availability for follow-up.

Exclusion Criteria:

* Patients refused to participate in the trial.
* Patients with any uncontrolled clinical disease (as evaluated by each patient's clinician), such as any associated rheumatologic, thyroid, cardiovascular, pulmonary, hematologic, or renal diseases, pregnancy, lactation, and neuropsychiatric disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in pain Scores as measured by the Visual Analog Scale | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Eman Khedr, MD, Principal Investigator — Professor of Neurology, Faculty of Medicine, Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khedr EM, Omran EAH, Ismail NM, El-Hammady DH, Goma SH, Kotb H, Galal H, Osman AM, Farghaly HSM, Karim AA, Ahmed GA. Effects of transcranial direct current stimulation on pain, mood and serum endorphin level in the treatment of fibromyalgia: A double blinded, randomized clinical trial. Brain Stimul. 2017 Sep-Oct;10(5):893-901. doi: 10.1016/j.brs.2017.06.006. Epub 2017 Jun 23. PMID 28684258